CLINICAL TRIAL: NCT03617003
Title: Phase I Study of WST11 Phototherapy for Upper Tract Urothelial Carcinoma
Brief Title: Treatment of Tumors in the Urinary Collecting System of the Kidney or Ureter Using a Light Activated Drug (WST11)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-140
Record Dates: First submitted 2018-08-01; First posted 2018-08-06 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Upper Tract Urothelial Carcinoma
Keywords: WST-11; Phototherapy; 18-140
MeSH Terms: interventions — Endoscopy

STUDY DESIGN:
Intervention Model Description: This a prospective, single institution, non-randomized open label phase 1 study.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- phototherapy with WST11 (Experimental): Patients with urothelial cancer that includes involvement of the upper urinary tract and have failed prior endoscopic treatment, refuse standard treatment, or are ineligible for curative surgical resection of the kidney or ureter will be offered WST11 VTP treatment to be provided at the time of scheduled endoscopic procedure. At the time of endoscopy, patients will be treated with VTP therapy applied to the site of the tumor.
  Interventions: Drug: WST11 mediated vascular targeted phototherapy (VTP); Procedure: Endoscopy

INTERVENTIONS:
Drug: WST11 mediated vascular targeted phototherapy (VTP) — All patients will receive intravenous administration of WST11 at a dose of 4 mg/kg, infused over 10 minutes while patients are under anesthesia during their endoscopy procedure, followed by immediate laser light application.
Procedure: Endoscopy — Endoscopy of the bladder

SUMMARY:
The purpose of this study is to test the safety of a combination of the study drug called WST11 and PDT. Photodynamic therapy (PDT) is a type of ablation therapy (treatment which destroys tumor cells) which has been previously approved for the treatment of patients with other cancers. It works by using a drug that is given through the vein and then is activated in the tumor by light administered during endoscopy, which results in destruction of the cancer cells.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older

  * Confirmed tissue diagnosis of urothelial carcinoma involving the ureter and/or renal pelvis with pathology reviewed at MSKCC
  * Residual or recurrent cancer following prior endoscopic treatment
  * Ineligible, unwilling or refusing to undergo surgical management by resection of involved kidney or ureter.
  * Karnofsky performance status ≥ 50%
  * Patients with existing ureteral obstruction and/or existing ureteral stent will be permitted. Demonstration of the site and degree of obstruction must be documented by retrograde pyelography at the time of initial and follow up endoscopic procedures within 60 days.
  * Patients should not have received any systemic therapy (including chemotherapy, biologic therapy or immunotherapy) ≤4 weeks prior to treatment
  * Patients on prophylactic or full-dose anticoagulation are eligible, provided the treating physician believes it is safe to temporarily withhold anticoagulation (see Section 9.2)
  * Adequate organ function defined at baseline as:

    * ANC ≥1,000/ µL
    * Platelets ≥75,000/ µL
    * Hb ≥9 g/dl
    * INR ≤1.5 (except for patients who are on full-dose warfarin)
    * Calculated creatinine clearance ≥40 ml/min (using Cockcroft-Gault method)
    * Total serum bilirubin ≤1.5 mg/dL
    * AST/ALT ≤5× upper limit of normal
  * Able to provide written informed consent

Exclusion Criteria:

* Pregnant or breast-feeding women. Women of childbearing potential (WOCBP) must undergo a negative pregnancy test (either serum or urine) prior to study entry. Both sexes must use contraception while on study. WOCBP include:

  * Any woman who has experienced menarche and who has not undergone surgical sterilization (hysterectomy, bilateral tubal ligation or oophorectomy) or who is not post-menopausal (defined as amenorrheic ≥12 consecutive months)
  * Women on hormone replacement therapy with documented serum follicle stimulating hormone level > 35 mIU/ml
  * Women who are using oral, implanted or injectable contraceptive hormones or mechanical products such as intrauterine device or barrier methods to prevent pregnancy or are practicing abstinence or where the partner is sterile
* T4 tumors with involvement of the bowel or major blood vessels • Any other medical or psychiatric comorbidities, including decompensated heart failure, unstable angina or coronary artery disease or severe pulmonary disease that, in the opinion of the study investigator, would make the patient a poor candidate for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2025-07-15 (Actual); Study Completion 2025-07-15 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated laser fluence rate | 2 years
  The MTD will be defined as the dose whose toxicity rate does not exceed an acceptable threshold of toxicity 20%.in this study, we shall start at 100mW/cm and will carefully escalate the dose to a maximum of 200 mW/cm.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Coleman, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm